CLINICAL TRIAL: NCT02974634
Title: Ostomy Telehealth For Cancer Survivors
Acronym: PCORI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: City of Hope Medical Center (Other); Yale University (Other); University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 826150
Record Dates: First submitted 2016-11-04; First posted 2016-11-28 (Estimated); Results first posted 2020-08-11 (Actual); Last update posted 2020-08-19 (Actual); Status verified 2020-08

CONDITIONS: Colostomy Stoma
Keywords: Ileostomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ostomy Self management Training (Active Comparator): Ostomy self-management Training group in which subject will learn using pouches and equipment, skin care, ostomy complications, nutritional needs, Impact on feelings, clothing changes, social relationships, being prepared for emergencies, Intimacy and sexuality, communication skills, tips for travelling and physical activity recommendations
  Interventions: Other: Ostomy self management training
- Usual care (Placebo Comparator): Usual care in peri-operative and long-term settings is not standardized for ostomy patients. Usual care does not provide any formal, reproducible training for patients or their caregivers. It typically consists of an Ostomy Care Nurse who works with patients and caregivers concerning technical issues (fitting, emptying, supplies, surrounding skin care, etc.) while the new ostomate is still an inpatient
  Interventions: Other: Ostomy self management training

INTERVENTIONS:
Other: Ostomy self management training — Ostomy Self management Training group in which subject will learn using pouches and equipment, skin care, ostomy complications, nutritional needs, Impact on feelings, clothing changes, social relationships, being prepared for emergencies, Intimacy and sexuality, communication skills, tips for travelling and physical activity recommendations

SUMMARY:
The purpose of this study is to test the benefits of an educational program, the Ostomy Self-Management Training (OSMT) program, for improving patient activation (preparedness to do self-care), self-efficacy (patients' ability to do self-care), knowledge of ostomy/urostomy self-care, quality of life, mood, use of medical services, and financial burden in patients with ostomies. The study will compare patients in the intervention (training) group and patients in the usual care group.

Subjects' participation in this study is expected to last about 7 months. The PI plans to enroll up to 176 subjects at 3 hospitals (University of Pennsylvania, Yale University School of Nursing, and City of Hope in Los Angeles). All patient telehealth education will be coordinated by the University of Arizona in Tucson, Arizona.

DETAILED DESCRIPTION:
Over one million individuals in the U.S. have ostomies. The American Cancer Society estimates 39,610 rectal cancer cases and 74,000 bladder cancer cases will be diagnosed in 2015. Of these, at least 30,000 will receive ostomies, and an additional unknown number due to gynecologic, other gastrointestinal tumors. The HRQOL impact is tremendous and greater than with many other cancer treatments. An ostomy is often a prolonged or lifelong disabling problem for cancer survivors. The adaptation period is quite variable. 18% of participants took at least one year, or never felt comfortable, in their ostomy care. Importantly, many patients cannot attend selfmanagement programs or patient groups for a myriad of reasons, including distance to travel, monetary outlays, comorbidities making travel difficult, or lack of access to transportation. In addition, a national shortage of OCNs means patients with an ostomy, whether newly placed or a long-term issue, receive little help.

It is imperative to study interventions for these cancer survivors aimed to limit family financial burdens, decrease medical care use, and improve well-being. This study has the potential to improve health care outcomes for cancer survivors with ostomies by enhancing their knowledge of and self-efficacy with ostomy care. This will be accomplished by improving the ability to communicate an established educational curriculum developed based on patient needs and desires and refined via a pilot study.

ELIGIBILITY:
Inclusion Criteria:

* All cancer survivors over 21 years of age having undergone a procedure that needed an intestinal stoma (fecal or urinary).

Exclusion Criteria:

* None

Ages: 21 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-08-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Krouse, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Penn Medicine, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Our Program Project team supports and promotes the sharing of resources as promoted by PCORI. Progress in medical research in general, and patient-reported outcome cancer research in particular, benefits from enhanced collaboration and sharing of data between productive, collaborative investigators. Based on this concept, our policy is to make the data collected as part of this proposal available to outside investigators based on the following guidelines.
  * Our final research data will be shared with interested colleagues through peer-reviewed publications and presentations at scientific meetings.
  * Any sharing of data with outside investigators must preserve the anonymity of the subjects per HIPAA guidelines.
  * Collaboration with key personnel identified in the proposal is encouraged, but not strictly required.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: July 2021.
Access Criteria: • All requests will be reviewed by the Principal Investigator and Co-Investigators named in this proposal who will apply the following principles when deciding whether the data should be shared:
  1. The request should be scientifically rigorous.
  2. If a collaboration with one or more project investigators is appropriate, such a collaboration should be established.
  3. The request should not conflict with ongoing or planned research by the PI or Co-Investigators.
  4. The request should not conflict with each institutional requirements. The investigators should agree to acknowledge the contribution in all presentations and publications.

REFERENCES:
- [Result] Sun V, Ercolano E, McCorkle R, Grant M, Wendel CS, Tallman NJ, Passero F, Raza S, Cidav Z, Holcomb M, Weinstein RS, Hornbrook MC, Krouse RS. Ostomy telehealth for cancer survivors: Design of the Ostomy Self-management Training (OSMT) randomized trial. Contemp Clin Trials. 2018 Jan;64:167-172. doi: 10.1016/j.cct.2017.10.008. Epub 2017 Oct 16. PMID 29051047
- [Result] Sun V, Bojorquez O, Grant M, Wendel CS, Weinstein R, Krouse RS. Cancer survivors' challenges with ostomy appliances and self-management: a qualitative analysis. Support Care Cancer. 2020 Apr;28(4):1551-1554. doi: 10.1007/s00520-019-05156-7. Epub 2019 Nov 13. PMID 31720825
- [Derived] Rock MC, Cidav Z, Sun V, Ercolano E, Hornbrook MC, Wendel CS, Mo J, Fellheimer H, McCorkle R, Holcomb M, Grant M, Weinstein RS, Krouse RS. Adapting to the burdens of care: a telehealth program for cancer survivors with ostomies. Support Care Cancer. 2022 Dec 14;31(1):15. doi: 10.1007/s00520-022-07461-0. PMID 36513895
- [Derived] Grant M, Sun V, Tallman NJ, Wendel CS, McCorkle R, Ercolano E, Simons C, Mo J, Raza S, Donahue D, Passero F, Henson J, MacDougall L, Friedlaender J, Pitcher P, Fry D, Yonsetto P, Holcomb MJ, Hornbrook MC, Weinstein RS, Krouse RS. Cancer survivors' greatest challenges of living with an ostomy: findings from the Ostomy Self-Management Telehealth (OSMT) randomized trial. Support Care Cancer. 2022 Feb;30(2):1139-1147. doi: 10.1007/s00520-021-06449-6. Epub 2021 Aug 26. PMID 34435212
- [Derived] Weinstein RS, Holcomb MJ, Mo J, Yonsetto P, Bojorquez O, Grant M, Wendel CS, Tallman NJ, Ercolano E, Cidav Z, Hornbrook MC, Sun V, McCorkle R, Krouse RS. An Ostomy Self-management Telehealth Intervention for Cancer Survivors: Technology-Related Findings From a Randomized Controlled Trial. J Med Internet Res. 2021 Sep 27;23(9):e26545. doi: 10.2196/26545. PMID 34086595
- See also: Cancer Survivors' Challenges With Ostomy Appliances and Self-Management: A Qualitative Analysis — https://pubmed.ncbi.nlm.nih.gov/31720825/
- See also: Ostomy Telehealth for Cancer Survivors: Design of the Ostomy Self-management Training (OSMT) Randomized Trial — https://pubmed.ncbi.nlm.nih.gov/29051047/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at three study sites through several mechanisms. These include identification of potential participants via institutional registry, records,databases.Referrals from site WOCNs, attending surgeons and other clinical providers; and through distribution of Institutional .
  Subjects were recruited from 11/01/16 to 10/01/2018.
Pre-assignment Details: All cancer survivors over 21 years of age who were at least six weeks after a surgical procedure that necessitated the creation of an intestinal stoma (fecal or urinary) were recruited. Survivors with temporary ostomies were included, and there was no maximum time since surgery.
Groups:
- Ostomy Self Management Training: The intervention arm integrates goal setting and problem-solving approaches to enhance buy-in and encourage ability to carry out ostomy self-care. The curriculum was delivered via four group sessions by trained ostomy certified nurses and peer/experienced ostomates. An additional session was offered to support persons to address their needs related to ostomy care. Telehealth real-time videoconferencing was used to enhance program delivery to participants, usually in their homes, in three different geographic areas across two time zones.
  Ostomy Self management Training group in which subject will learn using pouches and equipment, skin care, ostomy complications, nutritional needs, Impact on feelings, clothing changes, social relationships, being prepared for emergencies, Intimacy and sexuality, communication skills, tips for travelling and physical activity recommendations
- Usual Care: Patients in the usual care group receive regular ostomy care in a clinic or via email or phone, as well as a list of local and regional resources. These study subject were expected only to complete study surveys.
Period: Overall Study
Arm/Group | Ostomy Self Management Training | Usual Care
Started | 106 | 110
Completed | 78 | 89
Not Completed | 28 | 21
Not completed — Advanced disease | 12 | 3
Not completed — Noncompliance | 3 | 7
Not completed — intervention technology related issues | 5 | 0
Not completed — Death | 8 | 11

BASELINE CHARACTERISTICS:
Population: Study sites are three diverse geographic areas to ensure participation of diverse populations. Each of our participating institutions has a large catchment area which includes rural and inner-city populations. These are patient populations that are often under served as there is difficulty in participating in support groups or
Groups:
- Ostomy Self Management Training: Comparing OSMT group to UC group The intervention arm integrates goal setting and problem-solving approaches to enhance buy-in and encourage ability to carry out ostomy self-care. The curriculum was delivered via four group sessions by trained ostomy certified nurses and peer/experienced ostomates. An additional session was offered to support persons to address their needs related to ostomy care. Telehealth real-time videoconferencing was used to enhance program delivery to participants, usually in their homes, in three different geographic areas across two time zones.
  Ostomy Self management Training group in which subject will learn using pouches and equipment, skin care, ostomy complications, nutritional needs, Impact on feelings, clothing changes, social relationships, being prepared for emergencies, Intimacy and sexuality, communication skills, tips for travelling and physical activity recommendations
- Usual Care: Comparing OSMT group to UC group
  Subjects were provided with physician and Wound ostomy nurses contacts and written information about an ostomy care. These study subject were expected only to complete study surveys.
- Total: Total of all reporting groups
Arm/Group | Ostomy Self Management Training | Usual Care | Total
Number analyzed (Participants) | 106 | 110 | 216
Age, Continuous [Mean (Full Range); unit: years] | 61.6 [30 to 87] | 61.6 [33 to 92] | 61.6 [30 to 92]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 53 | 103
  Male | 56 | 57 | 113
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 8 | 20
  Not Hispanic or Latino | 94 | 102 | 196
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 6 | 3 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 7 | 17
  White | 76 | 90 | 166
  More than one race | 2 | 3 | 5
  Unknown or Not Reported | 11 | 7 | 18
Region of Enrollment [Number; unit: participants] — Research projects to be performed will include oversight of all aspects of the project including training and overseeing staff, participating in weekly conference calls, and coordinating data collection.The PIs will participate in data interpretation and dissemination of project findings.
  participants
    United States | 106 | 110 | 216

OUTCOME MEASURES:

1. Primary Outcome: Patient Activation Measure (PAM), a 100 Point Scale Determining Patient Engagement in Healthcare.
Description: The patient activation measure (PAM) is a 100-point, quantifiable scale determining patient engagement in healthcare. PAM uses a uni-dimensional, probabilistic Guttman-like scale that reflects a developmental model of activation involving four stages (see below). 0 indicates lower activation (worse) whereas 100 indicates higher activation (better)
  (1) believing the patient role is important, (2) having the confidence and knowledge necessary to take action, (3) actually taking action to maintain and improve one's health, and (4) staying the course even under stress.
Time Frame: baseline, on completion of session ( 5 weeks) and 6 month follow up
Population: Intent to treat participants who provided baseline and at least one followup measurement
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ostomy Self Management Training | Usual Care
Number analyzed (Participants) | 89 | 101
score on a scale
  Baseline: number analyzed (Participants) | 80 | 90
  Baseline | 66.9 (12.9) | 64.2 (15.8)
  Post session: number analyzed (Participants) | 82 | 90
  Post session | 67.6 (12.9) | 66.2 (13.5)
  6 months follow up: number analyzed (Participants) | 61 | 73
  6 months follow up | 70.7 (13.3) | 66.5 (12.3)
Statistical Analysis 1: Comparison: Ostomy Self Management Training vs Usual Care; Test type: Superiority; p = 0.06, t-test, 2 sided — Comparison of intervention and usual care at 6 month follow up; Slope = 1.04, 95% CI 2-sided [-3.5 to 5.6], Standard Error of Mean 2.32 — Interaction coefficient (slope) of arm by time period (6 months follow up vs baseline) from mixed linear model

2. Secondary Outcome: Self-Efficacy to Perform Ostomy Self-Management Behaviors
Description: Modified from Lorig and colleagues' Self-Efficacy to Perform Self-management Behaviors Scale, an outcome measure for Chronic Disease Management Interventions, this scale represents 8 domains with reported Cronbach's alpha for original scales: physical activity, information seeking,support, communication with HC providers, ostomy management , social and recreational, symptom management, and depression.
  Range 1 to 10, where higher is better outcome
Time Frame: baseline, on completion of session ( 5 weeks) and 6 month follow up
Population: Intent to treat participants who provided baseline and at least one followup measurement
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Ostomy Self Management Training: The intervention arm integrates goal setting and problem-solving approaches to enhance buy-in and encourage ability to carry out ostomy self-care. The curriculum was delivered via four group sessions by trained ostomy certified nurses and peer/experienced ostomates. An additional session was offered to support persons to address their needs related to ostomy care. Telehealth real-time videoconferencing was used to enhance program delivery to participants, usually in their homes, in three different geographic areas across two time zones. Self management Training group in which subject will learn using pouches and equipment, skin care, ostomy complications, nutritional needs, Impact on feelings, clothing changes, social relationships, being prepared for emergencies, Intimacy and sexuality, communication skills, tips for travelling and physical activity recommendations
Arm/Group | Ostomy Self Management Training | Usual Care
Number analyzed (Participants) | 89 | 101
score on a scale
  Baseline: number analyzed (Participants) | 86 | 99
  Baseline | 6.7 (2.1) | 7.0 (2.2)
  Post session: number analyzed (Participants) | 85 | 96
  Post session | 7.1 (2.0) | 7.3 (1.9)
  6 months follow up: number analyzed (Participants) | 66 | 79
  6 months follow up | 7.3 (2.2) | 7.1 (2.1)
Statistical Analysis 1: Comparison: Ostomy Self Management Training vs Usual Care; Test type: Superiority; p = 0.68, t-test, 2 sided — Comparison of intervention and usual care at 6 month follow up; Slope = 0.34, 95% CI 2-sided [-0.24 to 0.91], Standard Error of Mean 0.29 — Interaction coefficient (slope) of arm by time period (6 months follow up vs baseline) from mixed linear model

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the time subjects were part of the study from for 6 months.
Arm/Group | Ostomy Self Management Training | Usual Care
All-Cause Mortality (participants affected / at risk) | 8/106 | 11/110
Serious Adverse Events (participants affected / at risk) | 0/106 | 0/110
Other Adverse Events (participants affected / at risk) | 0/106 | 0/110

LIMITATIONS AND CAVEATS:
Randomization methods led to equal numbers of males and females,but did not achieve balance.Several intervention subjects completed surveys without attending sessions. Few participants dropped out of the study due to a technology related concern.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-11-06): https://cdn.clinicaltrials.gov/large-docs/34/NCT02974634/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-29): https://cdn.clinicaltrials.gov/large-docs/34/NCT02974634/SAP_001.pdf